CLINICAL TRIAL: NCT01164566
Title: Prospective Evaluation of Esophageal Pathology Treatment of Head and Neck Carcinoma
Brief Title: Esophagoscopy in Evaluating Treatment in Patients With Stage I-IV Head and Neck Cancer Who Are Undergoing Radiation Therapy and/or Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate Recruitment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00012541; NCI-2010-01466; CCCWFU 60110 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-07-07; First posted 2010-07-16 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Stage I Adenoid Cystic Carcinoma of the Oral Cavity; Stage I Mucoepidermoid Carcinoma of the Oral Cavity; Stage I Squamous Cell Carcinoma of the Hypopharynx; Stage I Squamous Cell Carcinoma of the Larynx; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Verrucous Carcinoma of the Larynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Adenoid Cystic Carcinoma of the Oral Cavity; Stage II Mucoepidermoid Carcinoma of the Oral Cavity; Stage II Squamous Cell Carcinoma of the Hypopharynx; Stage II Squamous Cell Carcinoma of the Larynx; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Verrucous Carcinoma of the Larynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): Patients undergo transnasal esophagoscopy at baseline and 3 months following completion of radiation therapy and/or chemotherapy.
  Interventions: Procedure: endoscopic procedure; Other: questionnaire administration

INTERVENTIONS:
Procedure: endoscopic procedure
  Other Names: endoscopy
Other: questionnaire administration — Ancillary studies

SUMMARY:
Brief Summary:

RATIONALE: Comparing results of diagnostic procedures, such as esophagoscopy, done before and after radiation therapy and/or chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This clinical trial is studying esophagoscopy in evaluating treatment in patients with stage I-IV head and neck cancer who are undergoing radiation therapy and/or chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess the prevalence of esophageal pathology (any esophageal abnormality, specifically: esophagitis, stricture/web, infections, neoplasms) as identified by esophagoscopy in patients with HNCA before and 3 months following primary radiation and/or chemotherapy.

II. To assess the changes in self-reported dysphagia symptoms as measured by the Eating Assessment Tool.

OUTLINE:

Patients undergo transnasal esophagoscopy at baseline and 3 months following completion of radiation therapy and/or chemotherapy.

ELIGIBILITY:
Inclusion

* Written informed consent must be obtained from all participants prior to beginning therapy; participants should have the ability to understand and be willing to sign a written informed consent document
* Primary diagnosis of head and neck carcinoma (oral, hypopharyngeal, laryngeal)
* Stage I-IV, undergoing treatment with radiation therapy +/- chemotherapy

Exclusion

* Medical history of esophageal dysfunction
* Pregnant women are not excluded from participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Abnormal endoscopic esophageal examination | 3 months following completion of radiation therapy
  Abnormal endoscopic esophageal examination, as defined by presence of: stricture, web, ring, erosive esophagitis, fungal esophagitis, viral esophagitis, Barrett's metaplasia, neoplasm, or other.

SECONDARY OUTCOMES:
Severity of self-rated swallowing dysfunction | 3 months following completion of radiation therapy
  Severity of self-rated swallowing dysfunction, as rated with the Eating Assessment Tool (0-40)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Rees, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States